CLINICAL TRIAL: NCT03359226
Title: Transcutaneous Submandibular Gland Biopsy: Feasibility of Repeat Biopsy as a Progression Marker for Parkinson&Apos;s Disease
Brief Title: Transcutaneous Submandibular Gland Biopsy: Feasibility of Repeat Biopsy as a Progression Marker for Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Charles Adler, Professor of Neurology, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-007240
Record Dates: First submitted 2017-11-14; First posted 2017-12-02 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Submandibular gland biopsy (Experimental): No treatment is being used in this study. Study participants will have bilateral submandibular gland biopsies.
  Interventions: Procedure: Submandibular gland biopsy

INTERVENTIONS:
Procedure: Submandibular gland biopsy — Needle biopsies of the right and left submandibular glands

SUMMARY:
The purpose of this study is to perform biopsies of one of the glands that make saliva. The biopsied tissue will then be analyzed to see if it has changes that occur in Parkinson's disease. This study will determine whether it is possible to do a second biopsy a few years after a previous biopsy and determine whether there are changes in the biopsy that would allow for analysis of disease progression.

DETAILED DESCRIPTION:
Tissue biopsies documenting the presence and density of Lewy type synucleinopathy (LTS) in living patients with probable Parkinsons disease (PD) would be extremely valuable as a diagnostic test, as a marker of molecular therapeutic target engagement and as a progression marker. Based on recent data from our group with both early and advanced PD patients, we propose to perform a second transcutaneous submandibular gland (SMG) needle core biopsy in 12 patients who have previously been biopsied and had LTS present in their SMG tissue.

ELIGIBILITY:
Inclusion criteria

1. PD patients ages up to age 85.
2. Previous participation in a SMG biopsy study at Mayo Clinic Arizona with a positive biopsy being reported

Exclusion criteria

1. Evidence for dementia that would preclude the patient from signing informed consent
2. History of bleeding diathesis or hematologic disorders
3. Medically unable to undergo a core needle biopsy of the submandibular gland
4. Prior treatment of the submandibular gland with botulinum toxin injections.
5. History of past or current acute infection or abscess of the submandibular gland.
6. History of past or current neoplastic process within the submandibular gland.
7. History of peripheral neuropathy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Presence of alpha-synuclein in the submandibular gland | baseline
  The biopsied submandibular gland tissue will be stained with an antibody for alpha-synuclein. The pathologist will review the slides and determine the number that show positive staining for neuronal elements. He will compare the number of positive slides between the right and left submandibular glands to see if they are similar.

CONTACTS AND LOCATIONS:
Overall Officials: Charles H Adler, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States